CLINICAL TRIAL: NCT05934149
Title: Lupus Nexus Landmark Study: A Prospective Registry and Biorepository
Brief Title: Lupus Landmark Study: A Prospective Registry and Biorepository
Status: Recruiting | Type: Observational
Sponsor: Lupus Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: LNX-Landmark-001
Record Dates: First submitted 2023-06-23; First posted 2023-07-06 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Systemic Lupus Erythematosus (SLE); Lupus Nephritis; Neuropsychiatric Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Lupus Vasculitis, Central Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood, blood derivatives, urine, stool, saliva, tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- New Onset: Individuals with a new diagnosis of SLE
- LN Active: Individuals with a recent diagnosis of Lupus Nephritis
- Extra-renal Flare: Individuals who have experienced a recent flare
- Prevalent: Individuals with lupus who do not meet the criteria for one of the other cohorts

SUMMARY:
The purpose of the registry and biorepository is to provide a mechanism to store clinical data, linked biospecimens and molecular data to support the conduct of future research on Systemic Lupus Erythematosus (SLE), including Lupus Nephritis (LN).

DETAILED DESCRIPTION:
This is a multicenter registry and biorepository conducted in the United States (US) and Canada. The registry will enroll over 3500 individuals with SLE over the course of five years into one of following four cohorts:

* New Onset: individuals with a new diagnosis of SLE
* Active Lupus Nephritis: individuals with a recent diagnosis of LN
* Extra-Renal Lupus Flare: individuals who have experienced a recent flare
* Prevalent Cases: individuals with lupus who do not meet the criteria for one of the other cohorts

The registry data will include but is not limited to: patient demographics, medical history, clinician-reported outcomes (ClinROs), patient-reported outcomes (PROs), social history and determinants of health, and environmental exposures. Participants will also be asked to allow access to their medical records.

Biological samples, including whole blood, urine, saliva, stool and tissue will be collected throughout the study. These biospecimens will be used for a broad range of analyses, including genetics, genomics, proteomics, biomarker discovery and microbiome profiling.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and comply with study procedures and voluntarily sign a written informed consent document
* Age 18 years or older at the time of enrollment
* Fulfill criteria for SLE based on one or more of the following classifications systems:

Systemic Lupus Erythematosus International Collaborating Clinic (SLICC) 2012 criteria; European Alliance of Associations for Rheumatology (EULAR)/American College of Rheumatology (ACR) 2019 criteria; 1997 revised ACR criteria; or Lupus is present per clinical assessment.

Exclusion Criteria:

* Not able to obtain consent
* Not able to meet protocol visit requirements
* Pregnant at the time of enrollment

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SLE
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Identify genetic drivers and antigenic targets, to elucidate mechanistic heterogeneity and correlate biomarkers to therapeutic responses. | up to 25 years
  Resource intended to be used to address research questions based upon three categorical time frames (historical, cross-sectional, and longitudinal) with specified scientific topics proposed upon request to access the resources.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Lim, MD, MPH, Principal Investigator — Emory University; Arezou Khosroshahi, MD, Principal Investigator — Emory University; Alfred Kim, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (21):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - Wallace Rheumatic Studies Center, Beverly Hills, California
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Massachusetts Memorial Health, Worcester, Massachusetts
  - Washington University, St Louis, Missouri
  - The Feinstein Institutes for Medical Research, Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - Northwell Health, New York, New York
  - SUNY Upstate, Syracuse, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - The MetroHealth System, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - University Health Network/Toronto Western Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and specimens may be provided to other researchers for additional research use.
Supporting Information: Study Protocol, ICF
Time Frame: Upon request, data and specimens may be made available after review by study team.
Access Criteria: The study team will review requests on an individual basis.